CLINICAL TRIAL: NCT05275179
Title: Pharmacokinetic of Intravenous Posaconazole in Critically Ill Patients
Brief Title: Pharmacokinetic of Posaconazole in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV7263
Record Dates: First submitted 2022-01-21; First posted 2022-03-11 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Therapeutic Drug Monitoring; Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Posaconazole Therapeutic Drug Monitoring: Therapeutic Drug Monitoring of posaconzole is performed by measuring posaconazole concentrations in serum
  Interventions: Other: Posaconazole Therapeutic Drug Monitoring

INTERVENTIONS:
Other: Posaconazole Therapeutic Drug Monitoring — Therapeutic Drug Monitoring is performed by measuring posaconazole concentrations in serum on seven consecutive days (anticipated).

SUMMARY:
The posaconazole pharmacokinetic in critically ill patients will be studied in a prospective, non-interventional, monocentric observational trial.

DETAILED DESCRIPTION:
The posaconazole pharmacokinetic in critically ill patients will be studied in a prospective, non-interventional, monocentric observational trial. Plasma specimens will be retrieved on consecutive days (max. 7 days) in order to measure posaconazole levels during the treatment episode.

ELIGIBILITY:
Inclusion Criteria:

* treatment with intravenous posaconazole
* critically ill patient
* written declaration of consent

Exclusion Criteria:

- no declaration of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients treated with posaconazole intravenously.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Posaconazole Drug Exposure | seven days from therapystart
  Measurement of posaconazole concentration in serum

SECONDARY OUTCOMES:
population-pharmacokinetic analysis 1 | 12 months after close out
  Analysis of Peak Plasma Concentration (Cmax) for posaconazole in the given cohort.
population-pharmacokinetic analysis 2 | 12 months after close out
  Analysis of Area under the plasma concentration versus time curve (AUC) for posaconazole in the given cohort.
Evaluation of probability of target attainment of posaconazole | 12 months after close out
  Analysis of Monte-Carlo-Simulations in order to asses novel dosing regimens for posaconazole.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Wichmann, Prof, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konig C, Gopfert M, Kluge S, Wichmann D. Posaconazole exposure in critically ill ICU patients: a need for action. Infection. 2023 Dec;51(6):1767-1772. doi: 10.1007/s15010-023-02078-9. Epub 2023 Jul 27. PMID 37498488